CLINICAL TRIAL: NCT03214692
Title: Potential Role of Gum Arabic as Antioxidant and Anti-inflammatory Agent in Hemodialysis Patients
Brief Title: Gum Arabic as Antioxidant and Anti-inflammatory in Hemodialysis Patients
Acronym: GA&CRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lamis Kaddam (Other)
Collaborators: Military Hospital Sudan (Unknown); University of Khartoum (Other)
Responsible Party: Sponsor-Investigator, Lamis Kaddam, Dr, Al-Neelain University
Organization: Al-Neelain University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA&CRF
Record Dates: First submitted 2017-06-18; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: End-Stage Renal Disease
Keywords: Gum Arabic; Renal failure; Hemodialysis; Antioxidant and anti-inflammatory
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Gum Arabic

STUDY DESIGN:
Intervention Model Description: Daily ingestion of Gum Arabic for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gum Arabic (Experimental): The patients will receive 30 grams of Gum Arabic dissolved in 200 ml of water to ingest orally
  Interventions: Dietary Supplement: Gum Arabic

INTERVENTIONS:
Dietary Supplement: Gum Arabic — Oral intake of GA in powder from30 grams per day

SUMMARY:
Oxidative processes increased in patients with renal failure and especially patients with end stage renal failure on dialysis. Oxidative stress plays a role in renal damage and also on cardiovascular disease, atherosclerosis, which can accelerate renal damage. Gum Arabic is claimed to have antioxidant effect and this will decrease the harmful effect of the free radical on patient on hemodialysis. In this study investigators are aiming to see the effect of Gum Arabic on Oxidative Stress and inflammatory markers in patients on regular hemodialysis.

DETAILED DESCRIPTION:
The oxidative stress reflects an imbalance between the systemic manifestation of reactive oxygen species and a biological system's ability to readily detoxify the reactive intermediates or to repair the resulting damage.

Cells continuously produce free radicals and reactive oxygen species (ROS) as part of metabolic processes. These free radicals are neutralized by an elaborate antioxidant defense system consisting of enzymes such as catalase, superoxide dismutase, glutathione peroxidase, and numerous non-enzymatic antioxidants, including vitamins A, E and C and glutathione.

Oxidative stress has been linked to the pathogenesis of a variety of diseases, such as renal disease, cardiovascular disease, atherosclerosis, hypertension, cancer, diabetes, arthritis neurodegenerative diseases (i.e., Alzheimer's and Parkinson's disease), and aging.

The prevalence and incidence of patient suffering from chronic renal failure is increasing worldwide and locally in Sudan(5). Several publication suggest that oxidative processes may be increased in patients with renal failure. As oxidative stress plays a role in renal damage it offers a potential target for therapeutic intervention.

There is a lot of factors that can lead to oxidative stress in patients with chronic kidney disease (CKD) . Intravenous administration of iron is widely prescribed in patients with chronic kidney disease (CKD) and can cause oxidative stress.Hemodialysis is often used for removal of excessive toxins, metabolic products, and blood components from patients with end-stage renal diseases (ESRD). Clinical studies have confirmed that hemodialysis (HD) is associated with the development of oxidative stress and disturbance in the enzyme systems that protect against oxygen free radicals.

The major cause of mortality in patients with end-stage renal failure receiving renal replacement therapy is cardiovascular disease . Cardiovascular disease (CVD) is the cause of death in 34% of hemodialysis (HD) patients. Increased lipid peroxidation and depletion of chain- breaking antioxidants may contribute to increased risk of atherosclerosis.

Antioxidants have been used as therapies to decrease oxidative stress and improve CVD risk in hemodialysis (HD) Patients .Many studies investigated the effects of antioxidant therapies on biomarkers of oxidative stress or clinical outcomes. The majority were small trials using a nonrandomized open-label design with a single HD group (no HD controls). The antioxidant used were Alpha-tocopherol , vitamin c decreased oxidative stress and N-acetylcysteine . N-acetylcysteine was the most efficacious agent. Others studies have used a combination of antioxidants that decreased oxidative stresses. Most of these intervention studies were done in HD patients .

Gum arabic is defined by the FAO/WHO Joint Expert Committee for Food Additives (JECFA) as 'a dried exudation obtained from the stems of Acacia Senegal tree or closely related species of Acacia (family Leguminosae).

GA is indigestible for both human and animals; Its fermentation by colonic intestinal bacteria leads to formation of various degradation products, such as short-chain fatty acids .Gum Arabic ingestion increases serum short chain fatty acid concentration, mainly butyrate and propionate. Serum butyrate concentration increased following administration of GA in healthy subjects. Oral intake of GA has been shown to provide several health benefits, such as prebiotic effects. GA significantly increases Bifidobacteria, Lactobacteria, and Bacteriodes in the gut. GA is claimed to have anti-cancer ,anti-malarial immune-modulatory and antioxidant effects. GA treatment has been shown to favorably influence clinical and laboratory results in rats with adenine-induced chronic renal failure CRF and in humans diagnosed with renal failure, reported that GA was able to decrease high levels of several pro-inflammatory cytokines in plasma and kidney of rats suffering from adenine-induced CRF.

The antioxidant effect of Gum Arabic has been observed in Number of published data .

More recently 2017 reported more evidence that GA has potent anti- oxidative effects in humans as demonstrated by its ability to increase TAC and to decrease oxidative stress markers in humans, Almost all previous studies were conducted in animal models or in vitro studies except the last one(17) . the increased intake of dietary antioxidants from GA may help to maintain an adequate antioxidant defense status . GA can be utilized in other clinical conditions and diseases caused by increased lipid peroxidation and tissue injury.

In this study investigators are aiming to see the effect of Gum Arabic on Oxidative Stress and inflammatory markers in patients on regular hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease patients on regular hemodialysis.

Exclusion Criteria:

* Patient known have ischemic heart disease (coronary artery disease),
* Pregnant women,
* Patient who have impaired liver function or hepatitis VIRUS positive,
* Patient who HIV positive and patient currently use of GUM Arabic.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Tumor necrosis factor alpha | Baseline and after 12 weeks
  pg/mL
Change from baseline Oxidative stress marker malondialdehyde | Baseline and after 12 weeks
  nmol/mL

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | Baseline and every four weeks for 12 weeks
  ml/ minute

CONTACTS AND LOCATIONS:
Locations (1):
- Military Hospital AlshaheedArif renal center, Khartoum, Umdorman, Sudan

REFERENCES:
- [Result] Kaddam L, Fadl-Elmula I, Eisawi OA, Abdelrazig HA, Salih MA, Lang F, Saeed AM. Gum Arabic as novel anti-oxidant agent in sickle cell anemia, phase II trial. BMC Hematol. 2017 Mar 16;17:4. doi: 10.1186/s12878-017-0075-y. eCollection 2017. PMID 28331623
- [Result] Ali BH, Al-Husseni I, Beegam S, Al-Shukaili A, Nemmar A, Schierling S, Queisser N, Schupp N. Effect of gum arabic on oxidative stress and inflammation in adenine-induced chronic renal failure in rats. PLoS One. 2013;8(2):e55242. doi: 10.1371/journal.pone.0055242. Epub 2013 Feb 1. PMID 23383316
- [Derived] Ali NE, Kaddam LA, Alkarib SY, Kaballo BG, Khalid SA, Higawee A, AbdElhabib A, AlaaAldeen A, Phillips AO, Saeed AM. Gum Arabic (Acacia Senegal) Augmented Total Antioxidant Capacity and Reduced C-Reactive Protein among Haemodialysis Patients in Phase II Trial. Int J Nephrol. 2020 Apr 9;2020:7214673. doi: 10.1155/2020/7214673. eCollection 2020. PMID 32328307